CLINICAL TRIAL: NCT06682819
Title: Metabolomics Analysis According to the Thickness of the Retinal Nerve Fiber Layer in Patients With NOHL Mutations
Brief Title: Metabolomics Analysis According to the Retinal Nerve Fiber Layer in Patients With NOHL Mutations (MétabOCT)
Acronym: MétabOCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Christophe Orssaud, Dr, Hôpital Necker-Enfants Malades
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MétabOCT-022022; 2022-A00537-36 (Other: ID-RCB)
Record Dates: First submitted 2024-10-30; First posted 2024-11-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects; Leber Hereditary Optic Neuropathy
Keywords: Leber hereditary optic neuropathy; Metabolomics analysis; OCT; mtDNA mutation
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Two arms will be constituted according to gender and crossed according to OCT data (Other): Considering the difference in NOHL prevalence in men and women, with a sex ratio of 7 men to 3 women, the metabolomic analysis data will be analyzed according to gender and OCT data.
  Interventions: Diagnostic Test: Optical coherent tomography

INTERVENTIONS:
Diagnostic Test: Optical coherent tomography — We compare the metabolomics profile of healthy patients based on the OCT appearance of the optic disc and RNFL

SUMMARY:
Leber hereditary optic neuropathy (LHON), due to mitochondrial DNA (mtDNA) mutations, is responsible for profound visual impairment. However, there is evidence that optic nerve damage begins before vision declines. There is no biomarker to determine when optic nerve damage begins before visual acuity decline occurs.

We hope that the analysis of metabolomics will reveal specific metabolomic profiles and different vitamin B3 and B9 levels depending on whether there are OCT signs of optic nerve damage in healthy patients with mtDNA mutations suggestive of LHON (11778, 3460 or 14484). The existence of an increase in the thickness of the optic fiber layer, whose normal values are well established, constitutes such a sign in favor of optic nerve damage.

DETAILED DESCRIPTION:
The primary objective is to determine the metabolomic profile of healthy patients carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with or without increased thickness of the optic fiber layer in OCT.

Given the difference in the prevalence of NOHL in men and women, with a sex ratio of 7 men to 3 women, this primary objective will be evaluated separately in these 2 groups of people.

Secondary objectives include Determination of the cellular metabolomic profile of healthy patients carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with or without increased thickness of the optic fiber layer in OCT.

Determination of the metabolomic profile in tears of healthy with an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with or without increased thickness of the optical fiber layer in OCT.

Comparison of the serum and cellular metabolomic profile of healthy with an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) according to the existence or not of an increase in thickness of the optical fiber layer in macular OCT and with a control population without mtDNA mutation; Determination of a different clinical and paraclinical (OCT) evolution according to the metabolomic profiles.

Determination of vitamin B3 and B9 levels of healthy with an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) according to the existence or not of an increase in the thickness of the optical fiber layer in macular OCT and with a control population without mtDNA mutation.

For the reasons mentioned above, the secondary objectives will be studied separately in men and women with the constitution of 2 groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with normal visual acuity and who has never had optic neuropathy, or Patient not carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with normal visual acuity and who has never had optic neuropathy;
* Patient agreeing to undergo an OCT;
* Patient agreeing to sign the informed consent;
* Patient affiliated to French social protection (Primary Health Insurance Fund, CMU, etc.) or European social protection.

Exclusion Criteria:

* Patient with or having had optic neuropathy regardless of its etiology
* Patient with glaucoma regardless of its etiology;
* Patient not wanting to undergo OCT;
* Patient not wanting to sign the informed consent;
* Patient not affiliated with French social protection (Primary Health Insurance Fund, CMU, etc.) or European.
* Patients less than 18 years old or over 60 years old
* Pregnant patient

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Metabolomic profile of healthy patients carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with or without increased thickness of the optic fiber layer in OCT | one year
  Results of the metabolomics analysis in the different groups established according to the appearance of the OCT and gender in healthy patients carrying mtDNA mutations suggestive of LHON (11778, 3460 or 14484).

SECONDARY OUTCOMES:
Metabolomic profile in tears of healthy patients carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with or without increased thickness of the optic fiber layer in OCT. | one year
  Results of the metabolome established on tears in the different groups established according to the appearance of the OCT and the gender in healthy patients carrying mtDNA mutation evocative of NOHL (11778, 3460 or 14484).
Cellular metabolomic profile of healthy patients carrying an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) with or without increased thickness of the optic fiber layer in OCT. | one day
  Results of the cellular metabolome established on leukocytes in the different groups established according to the appearance of the OCT and the gender in healthy patients carrying mtDNA mutation evocative of NOHL (11778, 3460 or 14484).
To assess a visual acuity evolution depending on the metabolomic profiles. | one year
  Monitoring of the clinical evolution of visual acuity for one year in the different groups established according to the OCT appearance and gender in healthy patients carrying mtDNA mutations suggestive of NOHL (11778, 3460 or 14484). comparison with metabolomic profiles.
To assess a different OCT evolution depending on the metabolomic profiles. | one year
  Monitoring of the evolution of visual acuity and OCT data for one year in the different groups established according to the OCT appearance and gender in healthy patients carrying mtDNA mutations suggestive of NOHL (11778, 3460 or 14484). comparison with metabolomic profiles.
Comparison of vitamin B3 and B9 levels in healthy patients with an mtDNA mutation suggestive of NOHL (11778, 3460 or 14484) according to macular OCT data and with a control population without mtDNA mutation. | one year
  Measurement of blood levels of vitamins B3 and B9 in different groups established according to OCT appearance and gender in healthy patients carrying mtDNA mutations suggestive of NOHL (11778, 3460 or 14484).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Orssaud, MD, Principal Investigator — Hopital Necker
Locations (1):
- HEGP, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No